CLINICAL TRIAL: NCT01306864
Title: Clinical Evaluation of Hemospray: Hemostasis of Active GI Luminal Tract Bleeding
Brief Title: Hemostasis of Active Gastrointestinal (GI) Luminal Tract Bleeding
Acronym: HALT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-017
Record Dates: First submitted 2011-02-17; First posted 2011-03-02 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Bleeding Peptic Ulcers
Keywords: Endoscopic Hemostasis; Peptic Ulcer; Recurrent Bleeding; Injection Therapy; Thermal Probe
MeSH Terms: conditions — Peptic Ulcer; Hemorrhage | interventions — Hemostasis, Endoscopic

ARMS (1):
- Hemospray Treatment (Experimental): Hemospray Kit
  Interventions: Device: Hemospray Kit

INTERVENTIONS:
Device: Hemospray Kit — Hemostasis of Arterial GI Bleeding
  Other Names: Endoscopic Hemostasis

SUMMARY:
The objective of this study is to show that Hemospray is effective in achieving initial hemostasis and documenting rate of further bleed when compared to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Bleeding peptic ulcer

Exclusion Criteria:

* Patient is: < 18 years of age
* Patient is unable to consent
* Patient is contraindicated to undergo endoscopy
* Patient has: coagulopathy, altered post surgical anatomy of the stomach, previously placed intrahepatic portosystemic shunt
* Patient is pregnant or lactating
* Patinet has an INR > 2.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-12; Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with further bleed | 72 Hours

SECONDARY OUTCOMES:
Proportion of patients with initial hemostasis | At the conclusion of the index procedure

CONTACTS AND LOCATIONS:
Locations (12):
- Canada (7):
  - Royal Alexandra, Edmonton, Alberta
  - Vancouver Coastal Health, Vancouver, British Columbia
  - Health Science Centre University of Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Center, London, Ontario
  - The Ottawa Hospital- Civic Campus and General Campus, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Erasmus MC University Medical Center, Rotterdam, Netherlands
- United Kingdom (3):
  - Belfast City Hospital, Belfast
  - Bradford Teaching Hospital NHS Foundation, Bradford
  - University of Nottingham, Nottingham

REFERENCES:
- [Derived] Sung JJY, Moreea S, Dhaliwal H, Moffatt DC, Ragunath K, Ponich T, Barkun AN, Kuipers EJ, Bailey R, Donnellan F, Wagner D, Sanborn K, Lau J. Use of topical mineral powder as monotherapy for treatment of active peptic ulcer bleeding. Gastrointest Endosc. 2022 Jul;96(1):28-35.e1. doi: 10.1016/j.gie.2022.01.020. Epub 2022 Feb 3. PMID 35124074